CLINICAL TRIAL: NCT03081208
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy and Safety of a Single Oral Administration of Nolasiban to Improve Pregnancy Rates Following IVF or ICSI in Day 3 and Day 5 Fresh Embryo Transfer Cycles
Brief Title: Phase 3 Placebo Controlled Study of Nolasiban to Improve Pregnancy Rates in Women Undergoing IVF/ICSI
Acronym: IMPLANT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-OBE001-005
Record Dates: First submitted 2017-03-06; First posted 2017-03-16 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Infertility
Keywords: IVF; ICSI
MeSH Terms: conditions — Infertility | interventions — nolasiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nolasiban 900 mg (Experimental)
  Interventions: Drug: Nolasiban 900mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nolasiban 900mg — Nolasiban dispersible tablets for single oral administration
  Arms: Nolasiban 900 mg
Drug: Placebo — Placebo dispersible tablets for single oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to confirm the efficacy of a single oral 900mg dose of nolasiban to increase the ongoing clinical pregnancy rate at 10 weeks post embryo transfer (ET) day.

DETAILED DESCRIPTION:
The study is a prospective, randomized, parallel group, double-blind, placebo-controlled study to confirm the efficacy and the safety of the oxytocin receptor antagonist, nolasiban, in 760 women undergoing fresh embryo transfer following in vitro fertilisation (IVF) or intra-cytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Key Inclusion Criteria:

* Indicated for IVF/ICSI in the context of assisted reproductive technology (ART)
* Follow a gonadotropin releasing hormone (GnRH) antagonist protocol, single injection of human chorionic gonadotropin (hCG) for triggering final follicular maturation and luteal phase support with vaginal micronized progesterone.
* Single, fresh D3 or D5 embryo transfer

Key Exclusion Criteria:

* Frozen-thawed embryo transfer
* More than 20 oocytes in the current controlled ovarian hyperstimulation (COH) cycle
* Serum P4 greater than 1.5 ng/mL on the day of hCG administration

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 810 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Intra-uterine pregnancy with fetal heart beat at 10 weeks | 10 weeks post ET day
  Intra-uterine pregnancy with fetal heart beat at 10 weeks post embryo transfer day

SECONDARY OUTCOMES:
Live birth | Up to 42 weeks of gestation
  Live birth after 24 weeks of gestation
Miscarriage | From 6 weeks post ET to 24 weeks gestation
  Any clinical pregnancy that does not result in a live birth prior 24 weeks
Intra-uterine pregnancy at 6 weeks | 6 weeks post ET
  Intra-uterine pregnancy with fetal heart beat at 6 weeks post ET day
Positive blood pregnancy test | 14 days post OPU
  Positive blood pregnancy test at 14 days post oocyte pick-up (OPU)

OTHER OUTCOMES:
Adverse events | Through study completion, up to 11 months
  Frequency and severity of treatment emergent adverse events
Neonatal assessments | Birth of infant until 28 days
  Incidence of any malformation or any significant morbidity during the neonatal period
ASQ-3 | 6 months after term
  Ages and Stages Questionnaire-3 (ASQ-3) domain score(s) at 6 months, adjusted for gestational age at birth

CONTACTS AND LOCATIONS:
Overall Officials: ObsEva SA, Study Director — Geneva
Locations (43):
- Belgium (4):
  - Investigator ID 1001, Brussels
  - Investigator ID 1002, Brussels
  - Investigator ID 1003, Brussels
  - Investigator ID 1004, Brussels
- Czechia (8):
  - Investigator ID 1107, Olomouc
  - Investigator ID 1101, Prague
  - Investigator ID 1102, Prague
  - Investigator ID 1103, Prague
  - Investigator ID 1104, Prague
  - Investigator ID 1108, Prague
  - Investigator ID 1109, Teplice
  - Investigator ID 1106, Zlín
- Denmark (4):
  - Investigator ID 1204, Copenhagen
  - Investigator ID 1205, Herlev
  - Investigator ID 1202, Hvidovre
  - Investigator ID 1203, Skive
- Estonia (2):
  - Investigator ID 1301, Tartu
  - Investigator ID 1303, Tartu
- Finland (3):
  - Investigator ID 1401, Helsinki
  - Investigator ID 1402, Helsinki
  - Investigator ID 1403, Oulu
- Germany (4):
  - Investigator ID 1501, Heidelberg
  - Investigator ID 1502, Lübeck
  - Investigator ID 1504, Mainz
  - Investigator ID 1503, Marburg
- Hungary (4):
  - Investigator ID 1601, Budapest
  - Investigator ID 1604, Budapest
  - Investigator ID 1603, Pécs
  - Investigator ID 1602, Tapolca
- Poland (6):
  - Investigator ID 1701, Bialystok
  - Investigator ID 1703, Bialystok
  - Investigator ID 1705, Bialystok
  - Investigator ID 1702, Katowice
  - Investigator ID 1704, Szczecin
  - Investigator ID 1706, Warsaw
- Spain (8):
  - Investigator ID 1801, Barakaldo
  - Investigator ID 1805, Barcelona
  - Investigator ID 1808, Barcelona
  - Investigator ID 1809, Leioa
  - Investigator ID 1804, Madrid
  - Investigator ID 1807, Madrid
  - Investigator ID 1811, Seville
  - Investigator ID 1806, Valencia

REFERENCES:
- [Derived] Griesinger G, Blockeel C, Pierzynski P, Tournaye H, Visnova H, Humberstone A, Terrill P, Pohl O, Garner E, Donnez J, Loumaye E. Effect of the oxytocin receptor antagonist nolasiban on pregnancy rates in women undergoing embryo transfer following IVF: analysis of three randomised clinical trials. Hum Reprod. 2021 Mar 18;36(4):1007-1020. doi: 10.1093/humrep/deaa369. PMID 33534895